CLINICAL TRIAL: NCT01267461
Title: Evaluation of the Proliferative Activities of Insulin Analogues in Primary Human Tumor Cells
Status: Available | Type: Expanded Access
Sponsor: Meir Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: 0015-10-MMC
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Endometrial Cancer; Colon Cancer
Keywords: To asses the biological actions of insulin analogs in primary tumor cells
MeSH Terms: conditions — Endometrial Neoplasms; Colonic Neoplasms

INTERVENTIONS:
Other: Tissue sample from tumor — Endometrial cancer specimens will be obtained from patients operated and treated at the Gynecologic Oncology Unit at Meir Medical Center. Colon cancer specimens will be obtained from patients that underwent colonoscopy at the Gastrointestinal Department at Meir Medical Center.

SUMMARY:
Recently the general medical literature has become aware that the use of certain long-acting insulin analogues could potentially increase cancer risk.During the last few years the investigators group generated information of both scientific and clinical relevance on the proliferative and anti-apoptotic actions of insulin analogues. The goal of this project is to evaluate the hypothesis that the proliferative and signalling activities elicited by insulin analogues may have a impact on tumor behavior. In this study the investigators will asses the biological actions of insulin analogs in primary tumor cells of endometrial and colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Endometrial and Colon Cancer

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult